CLINICAL TRIAL: NCT00777231
Title: Phase I/II Pilot Study of Mixed Chimerism to Treat Hemoglobinopathies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Talaris Therapeutics Inc. (Industry)
Collaborators: Duke University (Other); St. Christopher's Hospital for Children (Other); The Western Pennsylvania Hospital (Other); University of Florida (Other); Medical College of Pennsylvania Hospital (Other); Hahnemann University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICT-7621-042298; 549.02 (Other: SCX UofL IRB); 430.98 (Other: SC StC IRB); 445.98 (Other: NM UofL IRB); 417.98 (Other: AA WIRB); Pro00009281 (Other: SC DU IRB)
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell; Stem Cell; Tolerance; Bone Marrow Transplant; Total Body Irradiation (TBI); Apheresis; Aplastic Anemia; Hemoglobinopathies; Non Malignant
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia, Aplastic; Hemoglobinopathies

STUDY DESIGN:
Intervention Model Description: No control group used, single group for each of four different disease groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sickle Cell Disease (Experimental): Recipients treated with an enriched hematopoetic stem cell infusion
  Interventions: Biological: Enriched Hematopoetic Stem Cell Infusion
- Non-Malignant Disorders (Experimental): Recipients treated with an enriched hematopoetic stem cell infusion
  Interventions: Biological: Enriched Hematopoetic Stem Cell Infusion
- Aplastic Anemia (Experimental): Recipients treated with an enriched hematopoetic stem cell infusion
  Interventions: Biological: Enriched Hematopoetic Stem Cell Infusion
- Sickle Cell Disease : Extended Protocol (Experimental): Recipients treated with an enriched hematopoetic stem cell infusion and Campath 1H conditioning
  Interventions: Biological: Enriched Hematopoetic Stem Cell Infusion

INTERVENTIONS:
Biological: Enriched Hematopoetic Stem Cell Infusion — Enriched Hematopoetic Stem Cell Infusion

SUMMARY:
The goal of this research study is to establish chimerism and avoid graft-versus-host disease in patients with Hemoglobinopathies to halt disease progression.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is emerging as a therapeutic alternative for patients with sickle cell disease. Conventional HSCT therapy has been limited to extremely high-risk hemoglobinopathy patients. Those patients who may be difficult to identify before end-organ damage develops.

Also, conventional HSCT is only available to the minority of candidates who have Histocompatibility Leukocyte Antigen (HLA) identical siblings to donate bone marrow or mobilized peripheral blood stem cells.

This study proposes two important improvements over conventional HSCT:

* Donor peripheral blood or bone marrow will be processed via a new technology, which will deplete mature immune cells while enriching hematopoietic stem cells (HSC) and graft facilitating cells (FC).
* A reduced intensity recipient conditioning regimen will be used to promote mixed allogeneic chimerism, as opposed to full donor chimerism, following HSCT.

These two elements may significantly improve the benefit:risk ratio of HSCT for patients with hemoglobinopathies. Stem cell transplantation may become a more feasible option for patients that do not have HLA-identical siblings that can donate stem cells. Also, transplantation may be offered to patients earlier in the disease progression, before end-organ damage occurs.

ELIGIBILITY:
Inclusion Criteria:

The following criteria are established to identify subjects with sickle cell disease (SCD) who have a high predicted morbidity and are at risk for early mortality. Subjects with S/S disease, S/C disease, Hemoglobin H disease, Alpha Thalassemia Major, Thalassemia Major (also known as Cooley's anemia) or S/B* thalassemia and one or more of the following medical complications will be eligible:

* History of impaired neurological function and/or findings on Magnetic Resonance Image (MRI)/Magnetic Resonance Angiogram (MRA) that are associated with sickle cell disease
* More than 1 episode of acute chest syndrome with stage I or II pulmonary disease
* Osteonecrosis involving ≥ 2 joints
* Sickle cell nephropathy as evidenced by a glomerular filtration rate of 30% - 50% of the predicted normal
* Alloimmunization that is sufficient to interfere with the efficacy of chronic transfusion therapy
* Chronic or recurrent priapism
* Major visual impairment in one or both eyes with bilateral proliferative retinopathy
* Persistent disabling pain (≥ 2 episodes per year) despite trials of chronic transfusion and/or hydroxyurea at recommended doses for at least 6 months duration

Additional General Criteria:

Subjects must also meet all of the following general inclusion criteria:

* Subjects must have a related donor (identical or mismatched for 1, 2 or 3 HLA- A, HLA-B or HLA-DR loci).
* Subjects must have adequate cardiopulmonary function as documented by a left ventricular ejection fraction ≥ 50% (or within normal limits per Institutional criteria) or a left ventricular shortening fraction Within normal limits (WNL) per Institutional criteria, without inotropic support. If Ejection fraction is 40-50%, the patient may be considered for participation if cleared by a Cardiologist.
* Subjects must have adequate pulmonary function as documented by Diffusing capacity of the lung for carbon monoxide (DLCO) and Forced expiratory volume in 1 second (FEV1)

  * 50% predicted for age and size. If DLCO and FEV1 are between 40-50%, patient may be considered for participation if cleared by a Pulmonologist.
* Subjects must have adequate hepatic function as demonstrated by a serum albumin ≥ 3.0 mg/dL, and serum glutamic pyruvic transaminase (SGPT) or serum glutamic oxaloacetic transaminase (SGOT) ≤ 2.5 times the upper limit of normal.
* Subjects must have adequate renal function as demonstrated by a serum creatinine ≤ 1.5 mg/dL. If serum creatinine is ≥ 1.5 mg/dL, then a creatinine clearance test must be done and the result 50% of normal.
* Subjects or legal guardians must give written informed consent, and subjects must assent where age and intellectually appropriate.
* There are no age limits for this protocol.

Exclusion Criteria:

* Uncontrolled infection or severe concomitant diseases, which in the judgment of the Principal Investigator, could not tolerate transplantation.
* Severe impairment of functional performance as evidenced by a Karnofsky (patients ≥16 years old) or Lansky (children <16 years old) score <70%
* Stage III or IV sickle cell pulmonary disease
* Renal insufficiency (GFR < 25% of predicted normal for age)
* Subjects with a positive human immunodeficiency virus (HIV) antibody test result
* Subjects who are pregnant, as indicated by a positive serum human chorionic gonadotrophin (HCG) test
* Subjects of childbearing potential who are not practicing adequate contraception as defined by the investigator at the site
* Subjects must not have had previous radiation therapy that would preclude total body irradiation (as determined by a radiation oncologist).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-01; Primary Completion 2010-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Level of Donor Chimerism from Enriched Hematopoietic Stem Cell Engraftment | From one month to three years
  Tests are done at key time points to monitor for donor chimerism by evaluating presence of bone marrow-derived hematopoietic stem cells.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne T Ildstad, M.D., Study Director — Talaris Therapeutics Inc.
Locations (3):
- United States (3):
  - University of Louisville, Louisville, Kentucky
  - Duke University Medical Center, Durham, North Carolina
  - St. Christopher's Hospital for Children, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided